CLINICAL TRIAL: NCT03620942
Title: Development of Advanced Double Intravenous Vasopressor Automated (ADIVA) System With Improved Hemodynamic Trend Control During Spinal Anaesthesia for Caesarean Section
Brief Title: Development of Advanced Double Intravenous Vasopressor Automated (ADIVA) System
Acronym: ADIVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHF/CTG061/2017
Record Dates: First submitted 2018-08-05; First posted 2018-08-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hypotension; Anesthesia
Keywords: Maternal hypotension; Spinal anaesthesia; Caesarean section
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Vasoconstrictor Agents; Ephedrine

STUDY DESIGN:
Intervention Model Description: The first phase recruited 76 parturients. The second phase recruited 97 parturients. Parturients recruited from this phase will be randomized into either ADIVA group or DIVA group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADIVA system (Experimental): Vasopressor delivery automated system administering phenylephrine and ephedrine using a three-step algorithm vasopressor delivery technique
  Interventions: Drug: Phenylephrine; Drug: Ephedrine; Device: ADIVA System
- DIVA system (Active Comparator): Vasopressor delivery automated system administering phenylephrine and ephedrine using a two-step algorithm vasopressor delivery technique
  Interventions: Drug: Phenylephrine; Drug: Ephedrine; Device: DIVA System

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine will be administered with conditions as below:
  1. When systolic blood pressure is between 90-110% of baseline, 25mcg phenylephrine will be given either in infusion or bolus if heart rate ≥ 60 beats/min;
  2. When systolic blood pressure is less than 90% of baseline, 25 to 75mcg phenylephrine will be given either in infusion or bolus if heart rate ≥ 60 beats/min.
  Other Names: Vasopressor
Drug: Ephedrine — Ephedrine will be administered with conditions as below:
  1. When systolic blood pressure is between 90-110% of baseline, 2mg ephedrine will be given either in infusion or bolus if heart rate < 60 beats/min;
  2. When systolic blood pressure is less than 90% of baseline, 2 to 6mg ephedrine will be given either in infusion or bolus if heart rate < 60 beats/min.
  Other Names: Vasopressor
Device: ADIVA System — 1. When systolic blood pressure (SBP) is 100-110% of baseline, 25mcg phenylephrine (infusion) is given if heart rate ≥ 60 beats/min, and 2mg ephedrine (infusion) is given if heart rate < 60 beats/min;
  2. When SBP is 90-100% of baseline, 25mcg phenylephrine (infusion or bolus) is given if heart rate ≥ 60 beats/min, and 2mg ephedrine (infusion or bolus) is given if heart rate < 60 beats/min;
  3. When SBP is 80-90% of baseline, 50mcg phenylephrine (infusion or bolus) is given if heart rate ≥ 60 beats/min, and 4mg ephedrine (infusion or bolus) is given if heart rate < 60 beats/min;
  4. When SBP < 80% of baseline, 75mcg phenylephrine (infusion or bolus) is given if heart rate ≥ 60 beats/min, and 6mg ephedrine (infusion or bolus) is given if heart rate < 60 beats/min.
  Other Names: Advanced Double Intravenous Vasopressor Automated System
  Arms: ADIVA system
Device: DIVA System — DIVA system works as below:
  1. When systolic blood pressure is between 90 to 100% of baseline, 25mcg phenylephrine (bolus) will be given if heart rate ≥ 60 beats/min, whereas 2mg ephedrine (bolus) will be given if heart rate < 60 beats/min;
  2. When systolic blood pressure is less than 90% of baseline, 50mcg phenylephrine (infusion or bolus) will be given if heart rate ≥ 60 beats/min, whereas 4mg ephedrine (infusion or bolus) will be given if heart rate < 60 beats/min.
  Other Names: Double Intravenous Vasopressor Automated System
  Arms: DIVA system

SUMMARY:
Maternal hypotension during spinal anaesthesia for Caesarean delivery may bring various adverse effects. It is therefore important to closely monitor hypotension during spinal anaesthesia, however current technology does not allow the blood pressure monitoring to respond in timely manner should there be any occurrence of hypotension. The investigators developed an advanced double-intravenous vasopressor automated system (ADIVA) so as to tackle this issue via novel algorithm to control blood pressure more rigorously with more stable haemodynamic profiles.

DETAILED DESCRIPTION:
The incidence of maternal hypotension during spinal anaesthesia for Caesarean delivery is reported to be as high as 70-90%. The potential adverse effects resulting from maternal hypotension are nausea, vomiting, cardiac dysfunction, foetal acidosis and hypoxia.

Hypotension during spinal anaesthesia is currently detected using an intermittent blood pressure (BP) monitor cycling and reactive administration of vasopressors upon detection. The use of conventional non-invasive BP monitoring is limited by the time required to inflate and to deflate the cuffs commonly applied to the arm, which subsequently leads to a failure to react in a timely manner to BP changes when they occur.

The DIVA system (double-intravenous vasopressor automated system) previously developed helped tackle the limitations associated with the conventional management of hypotension in Caesarean sections under spinal anaesthesia. In a recent randomized controlled trial the DIVA system achieved less incidence of maternal hypotension compared to conventional management, however the side effects in mother and baby were still not fully eliminated.

In this proposed study a new algorithm for an advanced DIVA (ADIVA) system will be developed to control BP more rigorously by detecting BP with more stable haemodynamic profiles and thereby improve patient outcomes. The clinical trial will be conducted in 2 phases. The first phase included the use of ADIVA in 76 subjects who undergo spinal anaesthesia for Caesarean delivery to test its safety and efficacy. The second phase was a randomised controlled trial to investigate the use of ADIVA in comparison to the existing DIVA system in 97 patients undergoing spinal anaesthesia for Caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (American Society of Anesthesiologists physical status 1 and 2) parturients;
* With singleton full-term pregnancy;
* The indication for an elective cesarean delivery;
* The use of spinal anaesthesia for cesarean delivery;
* Anthropometric profile within the following range: age 21-50 years old, weight 40-90 kg and height of 145-170 cm.

Exclusion Criteria:

* Obstetric (e.g. pre-eclampsia, premature rupture of amniotic membranes for more than 48 hours, gestational diabetes on insulin, pregnancy-induced hypertension on medication) and uncontrolled medical (e.g. cardiac disease) complications;
* Contraindication to spinal anaesthesia and/or allergy to opioids.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female patients undergoing cesarean delivery will be recruited.
Enrollment: 173 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of events of Hypotension occurrence | 1 day (during cesarean delivery)
  Systolic blood pressure less than 80% of baseline systolic blood pressure

SECONDARY OUTCOMES:
Number of events of Hypertension occurrence | 1 day (during cesarean delivery)
  Systolic blood pressure more than 120% of baseline systolic blood pressure
Number of events of Nausea and vomiting occurrence | 1 day (during and after cesarean delivery)
  Nausea and vomiting during and after cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Singaraselvan Nagarajan, FCARCSI, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan HS, Nagarajan S, Chan JJI, Tan CW, Sultana R, Sia ATH, Sng BL. Evaluating an advanced double intravenous vasopressor automated system to treat hypotension during spinal anesthesia for cesarean delivery: a randomized controlled trial. BMC Anesthesiol. 2023 Jan 26;23(1):33. doi: 10.1186/s12871-023-01992-7. PMID 36703120
- [Derived] Nagarajan S, Chan JJI, Tan CW, Al-Hashim ZGA, Sultana R, Sia ATH, Sng BL. An advanced double intravenous vasopressor automated system to treat hypotension during spinal anaesthesia for caesarean section: A pilot study. Eur J Anaesthesiol. 2022 Jan 1;39(1):42-49. doi: 10.1097/EJA.0000000000001496. PMID 33831901

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT03620942/Prot_SAP_000.pdf